CLINICAL TRIAL: NCT05969730
Title: Efficacy and Safety of Baricitinib Versus Azathioprine in Combination With Topical Corticosteroids For Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Baricitinib Versus Azathioprine in Patients With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Malekan, Medical Intern, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.MAZUMS.REC.1402.17653
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Baricitinib; Azathioprine; Atopic Dermatitis; Moderate-to-Severe Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — baricitinib; Azathioprine

STUDY DESIGN:
Intervention Model Description: BAAZ-AD-IR is a single-center, open-label, randomized trial which will be conducted in Iran. Patients who meet eligibility criteria will randomize (1:1) to receive baricitinib 4 mg daily or azathioprine 1.5-2.5 mg/kg for 12 weeks. All patients will receive emollient daily. Four weeks prior to randomization, patients will discontinue tropical and systemic treatments for atopic dermatitis and will not be allowed to use them during the study. The drugs will be prescribed at visit 1 (randomization day, or four weeks after screening). All demographics and baseline information will be gathered at visit 1. Six weeks after visit 1, visit 2 will be scheduled for each patient. At visit 2, patients will be followed up. Twelve weeks after visit 1, visit 3 will be scheduled, and final assessments will be done.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Baricitinib 4-mg daily plus fluocinolone 0.025% topical ointment and daily emollient of urea 10% topical cream
  Interventions: Drug: Baricitinib 4 MG
- B (Experimental): Azathioprine 1.5-2.5 mg/kg plus fluocinolone 0.025% topical ointment and daily emollient of urea 10% topical cream
  Interventions: Drug: Azathioprine 1.5-2.5 mg/kg

INTERVENTIONS:
Drug: Baricitinib 4 MG — In visit 1 which will be scheduled after the washout period, demographic information and baseline assessment will be conducted and patients will randomize into arms, baricitinib 4-mg daily plus fluocinolone 0.025% topical ointment and daily emollient of urea 10% topical cream (Arm A). Six weeks after visit 1, Visit 2 will be set to follow up on the patient condition, particularly in terms of adverse effects, and reorder their intervention. Visit 3 will be 12 weeks after visit 1 to perform the final assessment.
  Arms: A
Drug: Azathioprine 1.5-2.5 mg/kg — In visit 1 which will be scheduled after the washout period, demographic information and baseline assessment will be conducted and patients will randomize into arms, azathioprine 1.5-2.5 mg/kg plus fluocinolone 0.025% topical ointment and daily emollient of urea 10% topical cream (Arm B). Six weeks after visit 1, Visit 2 will be set to follow up on the patient condition, particularly in terms of adverse effects, and reorder their intervention. Visit 3 will be 12 weeks after visit 1 to perform the final assessment.
  Arms: B

SUMMARY:
Atopic dermatitis, which is also known as atopic eczema, is a common inflammatory and chronic skin disease that is characterized by severe recurrent erythematous and pruritic lesions. Patients suffer from decreased quality of life and poor work productivity due to the disease complications like persistent scratching, skin pain, skin damage, sleep disturbances, and social/emotional distress. In the United States (US), the prevalence of adults with atopic dermatitis ranges from 5% to 10%.

The mainstay treatment for atopic dermatitis is emollient and tropical corticosteroids which could be efficient for less severe atopic dermatitis patients but moderate to severe patients usually need additional therapies like phototherapy or systemic medications.

It is revealed that Janus kinase signal transducers and activators of transcription (JAK-STAT) pathway has a prominent role in the development and progression of atopic dermatitis. JAK1/JAK2 inhibitor, baricitinib is a new-class orally available drug that is approved for systemic treatment of adult patients with moderate to severe atopic dermatitis. In the phase III clinical trial baricitinib 2-mg and 4-mg were shown efficient results as monotherapy of adult patients with moderate to severe atopic dermatitis who have an inadequate response to topical corticosteroids (TCS).

Azathioprine is an immunosuppressant and antimetabolite agent interferes with the formation of lymphocytes, and suppresses prostaglandin synthesis, both of which are implicated in the inflammation associated with eczema. Azathioprine can be used (off-label) for moderate to severe atopic dermatitis patients. Multiple studies have demonstrated that azathioprine might be effective for patients with moderate-to-severe atopic dermatitis. Azathioprine is usually prescribed when cyclosporine is either contraindicated or not effective.

This trial will be conducted to test the hypothesis that baricitinib 4-mg daily in combination with TCS is superior to azathioprine 1.5-2.5 mg/kg a day in combination with TCS for moderate-to-severe AD at week 12 in terms of efficacy and safety.

ELIGIBILITY:
Inclusion criteria

1. Patients with minimum age of 18 years and maximum 75 years at the time of informed consent
2. Patients who can read, understand, and provide written informed consent
3. Individuals with atopic dermatitis who have had a diagnosis for at least 12 months before to screening, as defined by the American Academy of Dermatology: Guidelines of care for the management of atopic dermatitis; Section 1. Diagnosis and assessment of atopic dermatitis [14].
4. Patients with moderate to severe atopic dermatitis which is defined as having Eczema Area and Severity Index (EASI) ≥ 16, validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) ≥ 3, and body surface area (BSA) affected ≥10%
5. Individuals who have a documented history of insufficient response to topical treatments (at least a moderate potency topical corticosteroids and/or cyclosporine for at least 4 weeks or the maximum duration recommended for the product prescribed) within the 6 months before screening determined by a dermatologist.
6. Patients who accept to discontinue using (1) oral systemic corticosteroids, (2) systemic immunomodulators such as methotrexate, cyclosporine, and mycophenolate mofetil, and (3) any other systemic therapy used to treat atopic dermatitis (approved or off-label use), for at least 4 weeks before randomization and throughout the study.
7. Patients who accept to discontinue (1) immune modulators (e.g., tacrolimus or pimecrolimus) (2) Topical phosphodiesterase type 4 (PDE-4) inhibitor (crisaborole) (3) sedating antihistamines (both old and new generations) (4) phototherapy, includes therapeutic phototherapy (psoralen plus ultraviolet A, ultraviolet B), excimer laser as well as self-treatment with tanning beds, at least 2 weeks prior to randomization.
8. Patients who agree to use emollients daily for at least 14 days before randomization and who agree to continue using emollients daily during the treatment period.
9. Patients undergoing chronic therapies to improve sleep should be on a stable dosage for at least 2 weeks before screening. Antihistamines with sedative effects are not approved.

Exclusion criteria

1. Patients who are currently suffering from or have a history of any concurrent skin disorders that would interfere with assessments of the study medication's effect on atopic dermatitis. For example, psoriasis or lupus erythematosus or eczema herpeticum, or erythrodermic, refractory, or unstable skin disease, including, but not limited, eczema that requires hospitalizations and/or intravenous treatment for skin infections.
2. Patients who have a known hypersensitivity to baricitinib or azathioprine or any component of these investigational products
3. Patients with any major concomitant disease that is expected to need the administration of systemic corticosteroids, such as unstable chronic asthma, or who otherwise interfere with trial participation or require active regular monitoring.
4. Patients who have been treated (1) Treatment with azathioprine in the previous 3 months (2) Having an experience of treatment with any oral JAK inhibitors including baricitinib < 4 weeks prior to randomization (3) Fusion proteins that target inflammatory pathways or monoclonal antibodies for less than 5 half-lives before randomization (4) Any parenteral corticosteroid administered by intramuscular/intravenous/intra-articular injection within 6 weeks before randomization or is anticipated to require a parenteral injection of corticosteroids during the study (5) probenecid at the time of randomization that cannot be discontinued for the duration of the study
5. Patients who have uncontrolled hypertension (repeated systolic blood Pressure >160 mmHg or diastolic blood pressure >100 mmHg) in a seated position.
6. Patients who have had any major surgery within 8 weeks before screening or will require major surgery during the study
7. Patients who are immunocompromised and have unacceptable risk for taking part in the trial.
8. Patients who have recently experienced myocardial infarction (MI) , or stroke, or venous thromboembolism (VTE) or recurrent VTE (≥2) , or unstable ischemic heart disease, or New York Heart Association Stage III/IV heart failure
9. Patients who have a history of or are currently suffering from any major and/or unstable disease that might provide an unacceptable risk while taking an investigational medication or interfere with data interpretation including but not limited mentally incompetent, current active pancreatitis, cardiovascular, endocrine, respiratory, gastrointestinal, hepatic, hematological, lymphoproliferative, neurological, or neuropsychiatric disorders.
10. Patients with a recent or present clinically significant viral, bacterial, fungal, or parasitic infection (including, but not limited, HIV, TB, Viral hepatitis)
11. Patients who have been exposed to a live vaccine 12 weeks before randomization, or are likely to require/receive a live vaccine throughout the course of the trial
12. Patients who have a history of persistent alcoholism, intravenous drug addiction, or other illicit substance usage during the last 2 years.
13. Patients who have a history of organ transplantation
14. Patients who have donated more than one unit of blood in the 4 weeks before screening or who intend to donate blood during the trial.
15. Patients who are Pregnant/lactating or planning to become pregnant during the study period (men and women)
16. Have any of the following specific abnormalities on screening laboratory tests:

    1. AST or ALT ≥2x upper limit of normal (ULN)
    2. Alkaline phosphatase (ALP) ≥2x ULN
    3. Total bilirubin ≥1.5x ULN
    4. Hemoglobin <10.0 g/dL (100.0 g/L)
    5. Total white blood cell count <2500 cells/μL (<2.50x103/μL or <2.50 GI/L)
    6. Neutropenia (absolute neutrophil count [ANC] <1200 cells/μL) (<1.20x103/μL or <1.20 GI/L)
    7. Lymphopenia (lymphocyte count <750 cells/μL) (<0.75x103/μL or <0.75 GI/L)
    8. Thrombocytopenia (platelets <100,000/μL) (<100x103/μL or <100 GI/L) i. eGFR <40 mL/min/1.73 m2 (Chronic Kidney Disease Epidemiology Collaboration equation [CKD-EPI] Creatinine 2009 equation).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | 12 weeks
  The EASI is used to measure extent of eczema in 4 body regions (head/neck, trunk, upper limbs, and lower limbs) and assesses the following 4 clinical signs: (1) Erythema/Redness, (2) Thickness/Edema/Papulation, (3) Excoriation/Scratching (4) Lichenification. The intensity of each sign in each body region is assessed as: none (0), mild (1), moderate (2) and severe (3). The EASI score is ranged from 0 to 72. The higher score indicates a worse condition.

SECONDARY OUTCOMES:
Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD) | 12 weeks
  The vIGA-AD showed the dermatologist's global assessment of the patient's overall severity of their atopic dermatitis based on a numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is taken to the degree of erythema, papulation/induration, oozing/crusting, and lichenification in patients. The higher score indicates a worse condition.
SCORing Atopic Dermatitis (SCORAD) | 12 weeks
  The SCORAD index measures 3 aspects of atopic dermatitis in patients and presents a general score (A/5 + 7*B/2 + C, maximum possible score of 103). These aspects include (A, 0-100%) the extent of disease with the rule of nines, (B, 0-18) disease severity through 6 clinical characteristics [(1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe)], and (C, 0-20) subjective symptoms of pruritus and sleep loss. The higher score indicates a worse condition.
Body surface area affected (BSA-Affected) | 12 weeks
  The SCORAD data will be used to calculate the body surface area affected by atopic dermatitis.
Dermatology Life Quality Index (DLQI) | 12 weeks
  The Dermatology Life Quality Index (DLQI) is a 10-item, validated, patient-administered quality-of-life questionnaire that includes six domains: symptoms and feelings, daily activities, leisure, job and school, personal relationships, and therapy. This scale's recall period is over the last week. Response categories include "not at all," "a little," "a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as 0. Total score vary from 0 to 30, with higher socre indicating a lower quality of life.
Itch Numeric Rating Scale (Itch NRS) | 12 weeks
  The Itch Numeric Rating Scale (Itch NRS) is an 11-point horizontal scale reported by the patient, ranging from 0 to 10, with 0 indicating "no itch" and 10 signifying "worst itch imaginable." Patients select the number that best describes the worst level of itching in the past 24 hours. The higher score indicates a worse condition.
Skin Pain Numeric Rating Scale (Skin Pain NRS) | 12 weeks
  The skin pain Numeric Rating Scale (skin pain NRS) is an 11-point horizontal scale reported by the patient, ranging from 0 to 10, with 0 indicating "no skin pain" and 10 signifying "worst skin pain imaginable." Patients select the number that best describes the worst level of skin pain in the past 24 hours. The higher score indicates a worse condition.
Atopic Dermatitis Sleep Scale (ADSS) | 12 weeks
  The Atopic Dermatitis Sleep Scale (ADSS) is a 3-item questionnaire, reported by patients and designed to measure the impact of itch on sleep including difficulty falling asleep, frequency of waking, and difficulty getting back to sleep over last night. Patients assess their difficulties falling asleep and going to sleep, items 1 and 3, respectively, using a 5-point Likert-type scale with responses ranging from 0 "not at all" to 4 "very difficult." In item 2. Patients indicate their frequency of waking up last night by choosing the number of times between 0 to 29. Each item is scored separately.
Patient-Oriented Eczema Measure (POEM) | 12 weeks
  The patient-oriented eczema measure (POEM) is a 7-item patient-reported questionnaire used to assess the severity of atopic dermatitis. Seven symptoms will be asked through questions including (itching, sleep disturbance, bleeding, weeping/oozing, cracking, flaking, and dryness/roughness) on a scale ranging from 0-4 (0=no days, 1=1-2 days, 2=3-4 days, 3=5-6 days, 4=everyday). Scores range from 0 to 28. The higher score indicates a worse condition.
Hospital Anxiety Depression Scale (HADS) | 12 weeks
  The Hospital Anxiety Depression Scale (HADS) is a patients-reported questionnaire with 14 items that evaluate a patient's degree of anxiety and depression during the previous week. Each item is scored on a 4-point scale, giving maximum scores of 21 for anxiety and depression.
Adverse Events (Safety assessment) | Throughout the study
  Investigators are responsible for appropriate medical care throughout the study and monitoring the all adverse effects of patients who have enrolled in this study. Also, investigators must document all related safety data as well as laboratory results based on the prepared guide/list below. The phone number of the responsible investigator will be available for each patient. The patients will be advised to inform the investigator about all unusual events they may experience. An in-person visit may be set for patients as needed.

CONTACTS AND LOCATIONS:
Locations (1):
- Iran, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Lio PA, Simpson EL, Han G, Soung J, Ball S, Sun L, Casillas M, DeLozier AM, Ding Y, Eichenfield LF. Improvement in sleep and itch and enhanced quality of life in adult patients with moderate-to-severe atopic dermatitis: results from a phase 3 trial of baricitinib therapy. J Dermatolog Treat. 2022 Jun;33(4):2057-2062. doi: 10.1080/09546634.2021.1914308. Epub 2021 Jun 28. PMID 34176407
- [Background] Simpson EL, Lacour JP, Spelman L, Galimberti R, Eichenfield LF, Bissonnette R, King BA, Thyssen JP, Silverberg JI, Bieber T, Kabashima K, Tsunemi Y, Costanzo A, Guttman-Yassky E, Beck LA, Janes JM, DeLozier AM, Gamalo M, Brinker DR, Cardillo T, Nunes FP, Paller AS, Wollenberg A, Reich K. Baricitinib in patients with moderate-to-severe atopic dermatitis and inadequate response to topical corticosteroids: results from two randomized monotherapy phase III trials. Br J Dermatol. 2020 Aug;183(2):242-255. doi: 10.1111/bjd.18898. Epub 2020 Mar 5. PMID 31995838
- [Background] Barbarot S, Auziere S, Gadkari A, Girolomoni G, Puig L, Simpson EL, Margolis DJ, de Bruin-Weller M, Eckert L. Epidemiology of atopic dermatitis in adults: Results from an international survey. Allergy. 2018 Jun;73(6):1284-1293. doi: 10.1111/all.13401. Epub 2018 Feb 13. PMID 29319189
- [Background] Wan H, Jia H, Xia T, Zhang D. Comparative efficacy and safety of abrocitinib, baricitinib, and upadacitinib for moderate-to-severe atopic dermatitis: A network meta-analysis. Dermatol Ther. 2022 Sep;35(9):e15636. doi: 10.1111/dth.15636. Epub 2022 Jul 27. PMID 35703351
- [Background] Wollenberg A, Nakahara T, Maari C, Peris K, Lio P, Augustin M, Silverberg JI, Rueda MJ, DeLozier AM, Pierce E, Yang FE, Sun L, Ball S, Tauber M, Paul C. Impact of baricitinib in combination with topical steroids on atopic dermatitis symptoms, quality of life and functioning in adult patients with moderate-to-severe atopic dermatitis from the BREEZE-AD7 Phase 3 randomized trial. J Eur Acad Dermatol Venereol. 2021 Jul;35(7):1543-1552. doi: 10.1111/jdv.17278. Epub 2021 Jun 5. PMID 33834521
- [Background] Bieber T, Reich K, Paul C, Tsunemi Y, Augustin M, Lacour JP, Ghislain PD, Dutronc Y, Liao R, Yang FE, Brinker D, DeLozier AM, Meskimen E, Janes JM, Eyerich K; BREEZE-AD4 study group. Efficacy and safety of baricitinib in combination with topical corticosteroids in patients with moderate-to-severe atopic dermatitis with inadequate response, intolerance or contraindication to ciclosporin: results from a randomized, placebo-controlled, phase III clinical trial (BREEZE-AD4). Br J Dermatol. 2022 Sep;187(3):338-352. doi: 10.1111/bjd.21630. Epub 2022 Jul 20. PMID 35484697
- [Background] Bracho-Borro M, Franco-Ruiz PA, Magana M. The use of azathioprine in atopic dermatitis: A review. Dermatol Ther. 2022 Sep;35(9):e15665. doi: 10.1111/dth.15665. Epub 2022 Jul 10. PMID 35751547
- [Background] Murphy LA, Atherton D. A retrospective evaluation of azathioprine in severe childhood atopic eczema, using thiopurine methyltransferase levels to exclude patients at high risk of myelosuppression. Br J Dermatol. 2002 Aug;147(2):308-15. doi: 10.1046/j.1365-2133.2002.04922.x. PMID 12174104
- [Background] Meggitt SJ, Gray JC, Reynolds NJ. Azathioprine dosed by thiopurine methyltransferase activity for moderate-to-severe atopic eczema: a double-blind, randomised controlled trial. Lancet. 2006 Mar 11;367(9513):839-46. doi: 10.1016/S0140-6736(06)68340-2. PMID 16530578
- [Background] Wollenberg A, Szepietowski J, Taieb A, Ring J. Corrigendum: Consensus-based European guidelines for treatment of atopic eczema (atopic dermatitis) in adults and children: part I. J Eur Acad Dermatol Venereol. 2019 Jul;33(7):1436. doi: 10.1111/jdv.15719. No abstract available. PMID 31259446
- [Background] Gerbens LAA, Hamann SAS, Brouwer MWD, Roekevisch E, Leeflang MMG, Spuls PI. Methotrexate and azathioprine for severe atopic dermatitis: a 5-year follow-up study of a randomized controlled trial. Br J Dermatol. 2018 Jun;178(6):1288-1296. doi: 10.1111/bjd.16240. Epub 2018 Apr 10. PMID 29237228
- [Background] Silverberg JI, Lei D, Yousaf M, Janmohamed SR, Vakharia PP, Chopra R, Chavda R, Gabriel S, Patel KR, Singam V, Kantor R, Hsu DY. What are the best endpoints for Eczema Area and Severity Index and Scoring Atopic Dermatitis in clinical practice? A prospective observational study. Br J Dermatol. 2021 May;184(5):888-895. doi: 10.1111/bjd.19457. Epub 2020 Sep 21. PMID 32959390
- [Background] Eichenfield LF, Tom WL, Chamlin SL, Feldman SR, Hanifin JM, Simpson EL, Berger TG, Bergman JN, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Krol A, Margolis DJ, Paller AS, Schwarzenberger K, Silverman RA, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 1. Diagnosis and assessment of atopic dermatitis. J Am Acad Dermatol. 2014 Feb;70(2):338-51. doi: 10.1016/j.jaad.2013.10.010. Epub 2013 Nov 27. PMID 24290431
- [Background] Reich K, Kabashima K, Peris K, Silverberg JI, Eichenfield LF, Bieber T, Kaszuba A, Kolodsick J, Yang FE, Gamalo M, Brinker DR, DeLozier AM, Janes JM, Nunes FP, Thyssen JP, Simpson EL. Efficacy and Safety of Baricitinib Combined With Topical Corticosteroids for Treatment of Moderate to Severe Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2020 Dec 1;156(12):1333-1343. doi: 10.1001/jamadermatol.2020.3260. PMID 33001140